CLINICAL TRIAL: NCT04925310
Title: IRIS - Infection With Respiratory Syncytial Virus in Infants - a Prospective Observational Cohort Study
Brief Title: Infection With Respiratory Syncytial Virus in Infants
Acronym: IRIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: MHH6309
Record Dates: First submitted 2021-05-20; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Respiratory Syncytial Virus Infections; Respiratory Syncytial Virus (RSV); Respiratory Syncytial Virus-bronchiolitis
Keywords: Respiratory Syncytial Virus (RSV); Infants; bronchiolitis; infection; cohort study
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Bronchiolitis; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Nasopharyngeal aspirate or swab for PCR pathogen screening Nasal fluid EDTA whole blood Serum Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RSV Bronchiolitis Group: hospitalized children with confirmed RSV infection between the first month of life and second year of life

SUMMARY:
IRIS (Infection with RespIratory Syncytial Virus) is an observational, multi-center study enrolling infants with severe RSV infection and healthy controls. Inclusion criteria are age below two years and hospitalization due to RSV infection at three German sites. Exclusion criteria are premature birth, congenital or acquired bronchopulmonary or cardiac diseases, and immunodeficiency. Blood and respiratory specimens are collected upon admission, and RSV and other pathogens are analyzed by multiplex polymerase chain reaction (PCR). Further biomaterials including plasma, nasal lining fluid, blood cells, DNA, and RNA specimens are sampled in a dedicated biobank. Detailed information on demographic characteristics and medical history is recorded, as well as comprehensive clinical data including vital signs, medication, and interventions.

DETAILED DESCRIPTION:
The IRIS study is designed as a multicentric, prospective, observational study initiated at Hannover Medical School, Germany. Upon enrollment, detailed data on demographic background, case histo-ry, clinical presentation, physical examination, diagnostic findings, treatment, and other patient related items is collected. Data on disease course, treatment, and complications is gathered. Blood and respiratory specimens are collected upon admission, and RSV and other pathogens are analyzed by multiplex polymerase chain reaction (PCR). Further biomaterials including plasma, nasal lining fluid, blood cells, DNA, and RNA specimens are sampled in a dedicated biobank (Hannover Unified Biobank). The study enrolls hospitalized children with confirmed RSV infection between the first month of life and second year of life. The diagnosis of RSV is evaluated by point-of-care testing (POCT, Sofia, Quidel, Kornwestheim, Germany), and positive findings are confirmed by polymerase chain reac-tion (PCR). Exclusion criteria are premature birth, congenital or acquired bronchopulmonary or car-diac diseases, and immunodeficiency. Healthy control probands are enrolled via recruitment of patients undergoing routine surgical procedures. Written informed consent is obtained from all parents and caregivers. Three local study centers in northern Germany (Hannover, Oldenburg, and Hildesheim) are contributing. All study sites are secondary or tertiary care hospitals and undergo extensive training in recruitment, biosample acquisition and processing, data collection and data entry, logistics, and security.

ELIGIBILITY:
Inclusion Criteria:

* RSV Infection, confirmed by polymerase chain reaction (PCR)
* Need for hospitalisation

Exclusion Criteria:

* premature birth
* bronchopulmonary diseases
* cardiac diseases
* immunodeficiency

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study enrolls hospitalized children with confirmed RSV infection between the first month of life and second year of life. The diagnosis of RSV is evaluated by point-of-care testing, and positive findings are confirmed by polymerase chain reac-tion (PCR). Exclusion criteria are premature birth, congenital or acquired bronchopulmonary or car-diac diseases, and immunodeficiency.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2013-10-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe RSV infection | 5 years
  Number of patients with severe RSV infection in three tertiary care centers in northern Germany.

SECONDARY OUTCOMES:
Outcome meassures of severe RSV infection in children (composite endpoint) | 5 years
  * length of hospitalisation (days)
  * length of additional oxygen supply (hours)
  * number of patients with need for intensive care treatment
  * number of patients with need for invasive ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Hansen Gesine, Prof, Principal Investigator — Hannover Medical School
Locations (2):
- Germany (2):
  - Hannover Medical School, Hanover, Lower Saxony
  - Universitätsklinik für Kinder- und Jugendmedizin Oldenburg, Oldenburg, Lower Saxony

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wetzke M, Funken D, Lange M, Bejo L, Haid S, Monteiro JGT, Schutz K, Happle C, Schulz TF, Seidenberg J, Pietschmann T, Hansen G. IRIS: Infection with RespIratory Syncytial Virus in infants-a prospective observational cohort study. BMC Pulm Med. 2022 Mar 15;22(1):88. doi: 10.1186/s12890-022-01842-1. PMID 35291998